CLINICAL TRIAL: NCT06381453
Title: Belimumab in the Management of Autoimmune Hepatitis: a Multi-centre, Open-label Trial of Add-on Belimumab Therapy to Standard of Care
Brief Title: Belimumab in Autoimmune Hepatitis
Acronym: BELief
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5037; 213168 (Other: Protocol Number)
Record Dates: First submitted 2024-02-29; First posted 2024-04-24 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Belimumab (Experimental): 200mg subcutaneous injection once a week
  Interventions: Drug: Belimumab Auto-Injector [Benlysta]

INTERVENTIONS:
Drug: Belimumab Auto-Injector [Benlysta] — Belimumab 200 MG/ML [Benlysta] will be given once a week as single-dose autoinjector
  Other Names: Benlysta

SUMMARY:
Background: Autoimmune hepatitis (AIH) is a rare chronic and lifelong liver disease. Untreated, disease progresses to end-stage cirrhosis and the focus of therapy is with immunosuppression. Current therapies are limited, not targeted, and associated with side effects that patients report reduce quality of life. AIH is believed to arise as a consequence of genetic & environmental risks. Disease is characterised by impaired immunoregulation, that favours a chronic and relapsing hepatitis. As well as recognising an important role for cytotoxic T cells and regulatory T cells, it has become apparent that in AIH, as well as other related autoimmune conditions, that B-cells are important. AIH is characterised by a plasma cell rich interface hepatitis and elevated IgG concentrations. Furthermore B-cell lineages interact with regulatory T-cells. Off-label use of Rituximab, an anti-CD20 agent, has been described for patients with AIH. A number of other ways of effectively targeting B-cells in the treatment of related autoimmune diseases have also been developed, but there have been limited studies in people living with autoimmune hepatitis. Belimumab is a human monoclonal antibody that inhibits B-cell activating factor (BAFF), also known as B-lymphocyte stimulator. It is approved in the Canada to treat systemic lupus erythematosus and lupus nephritis. It has not been studied before in AIH, but off-label reports are published. In an open-label clinical trial of people living with autoimmune hepatitis, the investigator will now formally study the effect of adding Belimumab to existing standard of care, with the goal being to evaluate treatment efficacy, the ability to reduce the burden of existing therapies whilst still controlling AIH disease, and to describe the tolerability & safety of Belimumab in people with AIH. Study Design: Open label, multi-centre, Canadian clinical trial. Patient population: Patients with autoimmune hepatitis, excluding patients with decompensated liver disease, who either have active disease despite standard of care (Group A), or who are maintained with disease remission using standard of care therapy (Group B). 48 patients will be recruited. Intervention: Weekly sub-cutaneous Belimumab. Duration: 72 weeks with interim analysis after 24 patients have been treated for 24 weeks; target recruitment 48 patients. Evaluation: Safety, Serum liver tests, quality of life, exploratory immunologic biomarkers, optional liver biopsy or fine needle liver aspirate. Primary end-point: Group A: 50% or more of subjects have an ALT<2x ULN & corticosteroids at a dose of </= 5mg of Prednisone (or equivalent); Group B: 50% or more of subjects able to maintain remission (normal ALT, normal IgG) on monotherapy with Belimumab. Conclusion: Using a combination of makers of treatment efficacy and safety the investigator will test the hypothesis that Belimumab should be further formally evaluated for people living with AIH.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Established clinical diagnosis of autoimmune hepatitis for at least 6 months
* Participant and clinician consent to follow AIH study therapy guidance for the duration of the open label clinical trial.

Group A:

* ALT > 2 x ULN in the absence of clinical evidence or concern for alternative etiology, and assessed by the investigator as related to active AIH using standard of care evaluation.
* Ongoing therapy with corticosteroids, and/or non-biologic immunosuppressants (AZA, MMF, MP) at a stable dosage for 4 weeks prior to screening

Group B:

* Patients with normal ALT and normal IgG concentration
* Ongoing therapy with single agent immunosuppression or immunosuppression with low dose Prednisone (10mg or less or budesonide 6mg or less)) alongside a second line agent (azathioprine, MMF, MP)
* Fibroscan showing liver stiffness of < 16kPa.

Exclusion Criteria:

* Primary liver disease other than AIH
* High probability of NAFLD as assessed by the investigator.
* ALT >10 x ULN
* Patients positive for HBsAg or HBcAb and/or Hepatitis C RNA
* Prior use if corticosteroid >15mg daily
* A positive pregnancy test and/or breast feeding
* The presence of advanced liver disease as defined by any of:

  1. Total Bilirubin >3 x ULN.
  2. Platelet count <100 x109/L.
  3. INR >1.5
* Live vaccines within 30 days prior to screening or at any time during the study
* The use of other biologics including TNF inhibitors, abatacept, or tocilizumab within the washout period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of treatment with Belimumab on AIH disease activity and corticosteroid use in the management of AIH | Week 48
  Group A:
  50% or more of subjects have an ALT<2x ULN and corticosteroids at a dose of </= 5mg of Prednisone (or equivalent).
  Group B:
  50% or more of subjects able to maintain remission (normal ALT, normal IgG) on monotherapy with Belimumab

SECONDARY OUTCOMES:
To investigate the effects of treatment with Belimumab on AIH disease activity and treatment burden | Week 48, Week 72
  * Proportion of subjects with ALT<2x ULN and able to stop corticosteroids
  * Proportion of patients with normal ALT, normal IgG and able to stop both corticosteroids and Azathioprine/Mycophenolate Mofetil/6-Mercaptopurine
  * Proportion of patients with normal ALT, normal IgG and able to stop corticosteroids
To measure the effects of treatment with Belimumab on AIH disease activity and treatment burden | Week 48, Week 72
  - Time to biochemical disease relapse (ALT>2xULN having reached values <2x ULN)
To see the effects of treatment with Belimumab on AIH disease activity and treatment burden | Week 48, Week 72
  * Changes in corticosteroid dose compared to baseline >/= 50% reduction
  * Changes in corticosteroid dose compared to baseline (expressed as % of initial dosage)
To measure the effects of Belimumab on markers of AIH disease activity | Week 24, Week 48, Week 72
  - Changes in serial biochemistry and IgG compared to baseline
To evaluate the effects of Belimumab on markers of AIH disease activity | Week 24, Week 48, Week 72
  - Changes in liver stiffness as measured by elastography compared to baseline
To outline the effects of Belimumab on Patient Reported Outcomes (PRO) | Week 24, Week 48, Week 72
  - Change in CLDQ domain scores from Baseline to end of treatment
To assess the effects of Belimumab on Patient Reported Outcomes (PRO) | Week 24, Week 48, Week 72
  - Change in Fatigue Scale domain scores from Baseline to end of treatment
To measure the effects of Belimumab on Patient Reported Outcomes (PRO) | Week 24, Week 48, Week 72
  - Change in SF-36 domain scores from Baseline to end of treatment
To evaluate the safety of Belimumab in patients with autoimmune hepatitis | Week 24, Week 48, Week 72
  - Incidence and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) from baseline to end of study.
To assess the safety of Belimumab in patients with autoimmune hepatitis | Week 24, Week 48, Week 72
  - Proportion of patients experiencing AE from baseline to end of study.
Safety and Tolerability | Week 24, Week 48, Week 72
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
To report the safety of Belimumab in patients with autoimmune hepatitis | Week 24, Week 48, Week 72
  - Change in suicidality score from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Hirschfield, MB BChir, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada